CLINICAL TRIAL: NCT02489981
Title: Specific Use-result Surveillance of Spiriva Respimat in Asthmatics (Patients With Severe Persistent Asthma)
Brief Title: Specific Use-result Surveillance of Spiriva Respimat in Asthmatics
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.525
Record Dates: First submitted 2015-05-21; First posted 2015-07-03 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Spiriva: Patients with severe persistent asthma
  Interventions: Drug: Spiriva

INTERVENTIONS:
Drug: Spiriva — 60 puffs

SUMMARY:
The safety of Spiriva® 2.5 µg Respimat® 60 puffs (hereinafter referred to as Spiriva® Respimat®) in patients with severe persistent asthma under the real-world use was not confirmed in clinical trials.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with severe persistent bronchial asthma
* Patient aged >= 15 years
* Patients who are naive to Spiriva Respimat and receive Spiriva Respimat for the first time for treatment of bronchial asthma on top of at least ICS (Inhaled corticosteroids) treatment.

Exclusion criteria:

* Patients who have a contraindication to Spiriva Respimat defined in the package insert for Spiriva Respimat
* Patients who have been enrolled this study before.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with severe asthma
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Hospital Felício Rocho, Belo Horizonte, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this Post Marketing Surveillance (PMS) was to investigate the safety and effectiveness of Spiriva Respimat in patients with severe persistent asthma under real-world use. This is a regulatory required PMS to investigate the safety and effectiveness of Spiriva® 2.5 μg Respimat® 60 puffs in patients.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Spiriva® Respimat®: Patients were administered Tiotropium as two puffs 2.5 microgram (μg) (5 μg total dose) via the Respimat inhaler once daily
Period: Overall Study
Arm/Group | Spiriva® Respimat®
Started (Started patients in the safety set) | 340
Completed | 213
Not Completed | 127
Not completed — Adverse Event | 21
Not completed — Insufficient effectiveness | 16
Not completed — Improved | 31
Not completed — Lost to Follow-up | 31
Not completed — Other than listed | 28

BASELINE CHARACTERISTICS:
Population: Safety set: This patient set includes all patients who were documented to have taken at least one dose of Spiriva Respimat except for patients who had no observation documented after entry, made invalid registration or were not under the appropriate site contact.
Arm/Group | Spiriva® Respimat®
Number analyzed (Participants) | 340
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: SafetySet
  Years | 60.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: Safety Set
  Participants
    Female | 183
    Male | 157
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Suspected Adverse Drug Reactions (ADRs)
Description: Percentage of patients with ADRs are presented. There was no primary outcome for effectiveness as the primary objective of the surveillance is the evaluation of safety.
Time Frame: Week 52
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Spiriva® Respimat®
Number analyzed (Participants) | 340
Percentage of participants | 5.59

2. Secondary Outcome: Change From Baseline in Asthma Control Status at Week 52
Description: The effectiveness was determined based on the change of asthma control status from baseline at Week 52 which is the secondary endpoint in the surveillance. The asthma control status was rated on a 3-point scale of well controlled, insufficiently controlled and poorly controlled based on asthma symptoms (in the daytime or at night), use of reliever and limitation of activities including exercise (based on "Asthma prevention and management guideline").
  Well-controlled=WC, Insufficiently-controlled=IC, Poorly-controlled=PC, Unknown=Unk, Missing=Miss, Baseline=BL, Week 52=W52
Time Frame: Baseline and Week 52
Population: Efficacy set: This patient set is a subset of the safety set that includes all patients in the safety set who have baseline and at least one available on-treatment asthma control status, Peak Expiratory Flow Rate (PEFR), Forced Expiratory Volume in one second (FEV1), Forced Vital Capacity (FVC) or Asthma Control Questionnaire (ACQ) 6 score.
Measure: Number; unit: Percentage of participants
Arm/Group | Spiriva® Respimat®
Number analyzed (Participants) | 248
Percentage of participants
  WC_BL & WC_52: number analyzed (Participants) | 12
  WC_BL & WC_52 | 66.67
  IC_BL & WC_52: number analyzed (Participants) | 117
  IC_BL & WC_52 | 58.12
  PC_BL & WC_52: number analyzed (Participants) | 111
  PC_BL & WC_52 | 35.14
  Unk_BL & WC_52: number analyzed (Participants) | 4
  Unk_BL & WC_52 | 50.00
  Miss_BL & WC_52: number analyzed (Participants) | 4
  Miss_BL & WC_52 | 0.00
  WC_BL & IC_52: number analyzed (Participants) | 12
  WC_BL & IC_52 | 0.00
  IC_BL & IC_52: number analyzed (Participants) | 117
  IC_BL & IC_52 | 17.95
  PC_BL & IC_52: number analyzed (Participants) | 111
  PC_BL & IC_52 | 22.52
  Unk_BL & IC_52: number analyzed (Participants) | 4
  Unk_BL & IC_52 | 25.00
  Miss_BL & IC_52: number analyzed (Participants) | 4
  Miss_BL & IC_52 | 25.00
  WC_BL & PC_52: number analyzed (Participants) | 12
  WC_BL & PC_52 | 0.00
  IC_BL & PC_52: number analyzed (Participants) | 117
  IC_BL & PC_52 | 4.27
  PC_BL & PC_52: number analyzed (Participants) | 111
  PC_BL & PC_52 | 17.12
  Unk_BL & PC_52: number analyzed (Participants) | 4
  Unk_BL & PC_52 | 0.00
  Miss_BL & PC_52: number analyzed (Participants) | 4
  Miss_BL & PC_52 | 0.00
  WC_BL & Unk_52: number analyzed (Participants) | 12
  WC_BL & Unk_52 | 0.00
  IC_BL & Unk_52: number analyzed (Participants) | 117
  IC_BL & Unk_52 | 2.56
  PC_BL & Unk_52: number analyzed (Participants) | 111
  PC_BL & Unk_52 | 0.90
  Unk_BL & Unk_52: number analyzed (Participants) | 4
  Unk_BL & Unk_52 | 25.00
  Miss_BL & Unk_52: number analyzed (Participants) | 4
  Miss_BL & Unk_52 | 0.00
  WC_BL & Miss_52: number analyzed (Participants) | 12
  WC_BL & Miss_52 | 33.33
  IC_BL & Miss_52: number analyzed (Participants) | 117
  IC_BL & Miss_52 | 17.09
  PC_BL & Miss_52: number analyzed (Participants) | 111
  PC_BL & Miss_52 | 24.32
  Unk_BL & Miss_52: number analyzed (Participants) | 4
  Unk_BL & Miss_52 | 0.00
  Miss_BL & Miss_52: number analyzed (Participants) | 4
  Miss_BL & Miss_52 | 75.00

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration.
Description: The safety set (The safety set includes all patients registered in the study and received the treatment) was used for adverse event reporting. A total of 359 patients were registered and Case Report Form (CRFs) were collected from 352 patients. The safety set includes 340 patients, excluding 12 patients who had no visit after registration.
Arm/Group | Spiriva® Respimat®
All-Cause Mortality (participants affected / at risk) | 1/340
Serious Adverse Events (participants affected / at risk) | 10/340
Other Adverse Events (participants affected / at risk) | 0/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva® Respimat® (N=340)
Anaphylactic reaction (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cerebral infarction (Nervous system disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Patients were not randomized and there are no within-study data. Patients in the study may differ from the overall asthma-treated population, or from treated patients who did not choose to participate in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02489981/SAP_000.pdf
  • Study Protocol (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT02489981/Prot_001.pdf